CLINICAL TRIAL: NCT06735963
Title: Evaluating the Impact of a Meta Quest 3 Gamified VR Rehabilitation Program on Pain, Functionality, Disability, and Balance in Knee Osteoarthritis: a Randomized Controlled Trial
Brief Title: Evaluating the Impact of a Meta Quest 3 Gamified VR Rehabilitation Program in Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Moayad Subahi, assistant professor, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAPO-02-K-012-2024-12-2379
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthristis
Keywords: osteoarthritis; virtual reality; game; rehabilitation
MeSH Terms: conditions — Osteoarthritis | interventions — Exercise; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional therapy control group (Active Comparator): The control group will receive conventional therapy alone, including exercises, ultrasound, and transcutaneous electrical nerve stimulation (TENS).
  Interventions: Procedure: Exercise; Device: Electrotherapy
- Experimental VR-based Group (Experimental): Experimental group receiving VR-based rehabilitation in addition to conventional physical therapy,
  Interventions: Device: Meta Quest 3 Virtual Reality; Procedure: Exercise; Device: Electrotherapy

INTERVENTIONS:
Device: Meta Quest 3 Virtual Reality — Immersive virtual reality Meta Quest 3 device
  Arms: Experimental VR-based Group
Procedure: Exercise — Traditional exercise program for knee OA patients
Device: Electrotherapy — Electrotherapy including Therapeutic Ultrasound (US) and Transcutaneous Electrical Nerve Stimulation (TENS)

SUMMARY:
The goal of this clinical trial is to learn if a gamified virtual reality (VR) rehabilitation program can effectively reduce pain, improve functionality, and enhance balance in adults aged 40-64 years diagnosed with knee osteoarthritis. The main questions it aims to answer are:

Can the VR rehabilitation program reduce pain and disability compared to conventional physical therapy alone? Can the VR rehabilitation program improve balance and functionality in patients with knee osteoarthritis? Researchers will compare a group receiving the VR-based rehabilitation program alongside conventional therapy to a group receiving only conventional therapy to see if the addition of VR leads to superior outcomes.

Participants will:

Undergo either VR-based rehabilitation combined with conventional therapy or conventional therapy alone.

Complete assessments at three time points (baseline, 3 weeks, and 7 weeks) using measures such as pain scales, disability indices, and balance tests.

DETAILED DESCRIPTION:
This randomized controlled trial will evaluate the impact of a gamified virtual reality (VR) rehabilitation program using the Meta Quest 3 device on pain, functionality, disability, and balance in individuals with knee osteoarthritis (OA). The study aims to address the limitations of traditional physical therapy by integrating immersive and engaging VR exercises to enhance patient adherence and therapeutic outcomes.

Eligible participants will be adults aged 40-64 years diagnosed with stage 2 or 3 knee OA based on the American College of Rheumatology criteria. Participants will be randomized into two groups: an experimental group receiving VR-based rehabilitation in addition to conventional physical therapy, and a control group receiving only conventional therapy. Both groups will undergo a 3-week intervention, consisting of 15 sessions conducted five times weekly.

The experimental group will use the Meta Quest 3 VR device for a gamified exercise program, incorporating two key modules:

Fruit Ninja VR - This module will focus on upper and lower body coordination, proprioception, and reaction time through interactive slicing motions.

PowerBeats VR - This module will emphasize endurance, knee stability, and functional coordination via rhythm-based punching and dodging activities.

Both modules are designed to engage participants in dynamic movements that promote balance, proprioception, and functional stability, tailored to address the needs of individuals with knee OA. The control group will receive conventional therapy alone, including exercises, ultrasound, and transcutaneous electrical nerve stimulation (TENS).

Outcome measures will be assessed at baseline, immediately post-intervention (3 weeks), and at follow-up (7 weeks). These include:

Pain: Visual Analog Scale (VAS) Functionality: Six-Minute Walk Test (6MWT) Disability: Western Ontario and McMaster Universities Arthritis Index (WOMAC) Balance: Berg Balance Scale (BBS) The trial hypothesizes that the experimental group will demonstrate superior improvements in pain, functionality, disability, and balance compared to the control group. Statistical analyses will include repeated measures ANOVA to assess differences across time points and between groups.

Ethical approval has been obtained from the Umm Al-Qura University Biomedical Research Ethics Committee, and informed consent will be secured from all participants before participation. This study aims to contribute to the growing body of evidence supporting the integration of VR technologies into rehabilitation practices, particularly for musculoskeletal conditions like knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-64 years
* Diagnosis: Knee OA (Stages 2 or 3 based on American College of Rheumatology criteria)
* Ability to read and understand Arabic

Exclusion Criteria:

* Recent lower extremity surgery/fractures
* Other rheumatologic or cardiovascular conditions
* Visual/auditory impairments
* Dizziness or vertigo

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-11 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Pain | From enrolment to the end of treatment at 7 weeks
  Visual Analog Scale (VAS)
Function | From enrolment to the end of treatment at 7 weeks
  six-Minute Walk Test (6MWT)
Disability | From enrolment to the end of treatment at 7 weeks
  Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Balance | From enrolment to the end of treatment at 7 weeks
  Berg Balance Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Umm Al-Qura University, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiani S, Rezaei I, Abasi S, Zakerabasali S, Yazdani A. Technical aspects of virtual augmented reality-based rehabilitation systems for musculoskeletal disorders of the lower limbs: a systematic review. BMC Musculoskelet Disord. 2023 Jan 3;24(1):4. doi: 10.1186/s12891-022-06062-6. PMID 36597077
- [Background] Stanica IC, Moldoveanu F, Portelli GP, Dascalu MI, Moldoveanu A, Ristea MG. Flexible Virtual Reality System for Neurorehabilitation and Quality of Life Improvement. Sensors (Basel). 2020 Oct 23;20(21):6045. doi: 10.3390/s20216045. PMID 33114272
- [Background] Blasco J, Igual-Camacho C, Blasco M, Anton-Anton V, Ortiz-Llueca L, Roig-Casasus S. The efficacy of virtual reality tools for total knee replacement rehabilitation: A systematic review. Physiother Theory Pract. 2021 Jun;37(6):682-692. doi: 10.1080/09593985.2019.1641865. Epub 2019 Jul 17. PMID 31313607